CLINICAL TRIAL: NCT03573895
Title: Comparison of Acute Effects of Stretching and Foam-rolling
Brief Title: Stretching vs Foam-rolling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Albert Pérez Bellmunt, Director, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P2/02
Record Dates: First submitted 2018-06-19; First posted 2018-06-29 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Muscle Relaxation
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Foam-Roller (Experimental)
  Interventions: Other: Foam-Roller
- Neuromuscular Stretching (Experimental)
  Interventions: Other: Neuromuscular stretching
- Pasive stretching (Experimental)
  Interventions: Other: Pasive stretching
- Control (No Intervention)

INTERVENTIONS:
Other: Foam-Roller — Application of foam roller in the posterior part of thigh.
  Arms: Foam-Roller
Other: Neuromuscular stretching — Use of a neuromuscular stretching applied to the hamstring muscles
  Arms: Neuromuscular Stretching
Other: Pasive stretching — Use of a pasive stretching applied to the hamstring muscles
  Arms: Pasive stretching

SUMMARY:
The study aims to compare the acute effects of the aplication of foam-rolling and stretching over the hamstrings flexibility.

The secondary objective is to determine which time can permit the obtention of better results.

ELIGIBILITY:
Exclusion Criteria:

* Pregnant women
* Musculoskeletal disorder in the last 3 months
* Surgical interventions in lower limbs in the last 6 months
* Psychological or nervous alterations
* Uncomprehension of the indications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Hamstring flexibility change | 0 seconds, 30 seconds and 2 minutes
  Measurement of the hamstring muscles flexibility change by the use of the Sit-and-Reach test

SECONDARY OUTCOMES:
Triceps surae flexibility change | 0 seconds, 30 seconds and 2 minutes
  Measurement of the triceps surae flexibility change by the use of the Lunge test
Fatigue perception | 0 seconds, 30 seconds and 2 minutes
  Measurement of the fatigue sensation by the use of the Modified Borg Scale

CONTACTS AND LOCATIONS:
Overall Officials: Albert Pérez-Bellmunt, PhD, Principal Investigator — Anatomy lecturer
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided